CLINICAL TRIAL: NCT02388295
Title: A 12-Week, Multicenter, Randomized, Parallel-Group Study to Assess the Safety, Tolerability, Pharmacokinetics, Biomarker Effects, Efficacy, and Effect on Microglia Activation, as Measured by Positron Emission Tomography, of AZD3241 in Subjects With Multiple System Atrophy
Brief Title: AZD3241 PET MSA Trial, Phase 2, Randomized,12 Week Safety and Tolerability Trial With PET in MSA Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0490C00023
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-07

CONDITIONS: Multiple System Atrophy, MSA
Keywords: Multiple System Atrophy (MSA), PET imaging, myeloperoxidase (MPO) inhibitor
MeSH Terms: conditions — Multiple System Atrophy; Thyroid Dyshormonogenesis 2A | interventions — AZD3241

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZD3241 (Experimental): Subjects will be randomized to one of the two doses of AZD3241 or placebo in a 1:1:1 ratio.
  Interventions: Drug: AZD3241
- Placebo to match AZD3241 (Placebo Comparator): Subjects will be randomized to one of the two doses of AZD3241 or placebo in a 1:1:1 ratio.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD3241 — Drug: AZD3241 administered for 12 weeks orally as a tablet.
  Other Names: AZD3241 to match placebo administered for 12 weeks.
  Arms: AZD3241
Drug: Placebo — Placebo to match AZD3241 administered for 12 weeks orally as a tablet.
  Other Names: Placebo to match AZD3241 administered for 12 weeks.
  Arms: Placebo to match AZD3241

SUMMARY:
AZD3241 myeloperoxidase (MPO) inhibitor trial is assessing safety and tolerability, randomized trial, in patients with Multiple System Atrophy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 30-80 years, inclusive, at screen.
2. Meet criteria for diagnosis of probable or possible MSA according to the consensus criteria (Gilman et al. 2008 ).
3. "High-affinity binder" or "mixed-affinity binder" for TSPO, as confirmed by prospective genotyping of TSPO polymorphism during screen.
4. Subjects must understand the nature of the study and must provide signed and dated written informed consent in accordance with local regulations before the conduct of any study-related procedures. The informed consent should reflect the protocol stipulations concerning the use of contraception.
5. Medical treatment of MSA and co-morbid medical conditions must be stable for at least 30 days prior to screen and between screen and baseline.
6. Written and oral fluency in the local language.
7. Able and willing to participate in all scheduled evaluations, abide by all study restrictions, and complete all required tests and procedures.
8. In the opinion of the investigator, the subject must be considered likely to comply with the study protocol and to have a high probability of completing the study.
9. Able to swallow tablets whole.

Exclusion Criteria:

1. Prior participation in any AZD3241 study.
2. Magnetic resonance imaging (MRI) performed during screen not consistent with diagnosis of MSA.
3. Received a PET scan within the last 12 months.
4. Negative Allen test in both hands, unless the brachial artery is used for arterial cannulation.
5. Subjects determined to be "low affinity binders" by TSPO genotyping.
6. Claustrophobia that would contraindicate a brain MRI scan or brain PET scan.
7. Pregnancy, lactation, or, if female of childbearing potential, positive serum β-hCG at screen or positive urine β-hCG at baseline (Day -1).
8. Initiation or change in pharmacologic therapy for symptoms of MSA within 30 days prior to screen or between screen and baseline (Day -1).
9. Significant neurological disease affecting the central nervous system (CNS), other than MSA
10. History of brain surgery for parkinsonism.
11. History of stem cell treatment.
12. Seizure disorder, unless well controlled and for which treatment has been stable for at least 30 days prior to screen and between screen and baseline (Day -1).
13. Presence of any clinically significant medical condition
14. History or presence of thyroid disease.
15. Any abnormal TSH or Free T4 test result at screen or baseline (Day -1).
16. History or presence of gastrointestinal disorders or other disease known to interfere with absorption, distribution, metabolism or excretion of drugs
17. History or presence of renal disease or impaired renal function.
18. A QT interval corrected according to the Fridericia procedure (QTcF) interval measurement > 450 msec at screen (single ECG) or baseline (Day -1) (mean of three ECG measurements) or a family history of long-QT syndrome.
19. Uncontrolled hypertension
20. History or presence of diabetes, unless glucose levels have been well controlled and for which treatment has been stable for at least 30 days prior to screen and between screen and baseline (Day -1).
21. History of cancer within the last 5 years, with the exception of nonmetastatic basal cell carcinoma of the skin.
22. Any clinically important abnormality, as determined by the investigator, on physical examination or vital signs, ECG, or clinical laboratory test results other than abnormality due to a stable, well-controlled medical condition; or any abnormality that could be detrimental to the subject or could compromise the study.
23. Use of potent inhibitors of CYP3A4, Use of potent inducers of CYP3A4 and/or Use of drugs mainly metabolized by CYP3A4
24. Treatment with any investigational drug or device within 60 days or five half-lives prior to screen, whichever is longer, or between screen and baseline (Day -1).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2016-09-19 (Actual); Study Completion 2016-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (7):
  - Research Site, Stanford, California
  - Research Site, New Haven, Connecticut
  - Research Site, Tampa, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, New York, New York
- Research Site, Innsbruck, Austria
- Research Site, Turku, Finland
- France (2):
  - Research Site, Bordeaux
  - Research Site, Toulouse
- Research Site, Salerno, Italy
- Research Site, Stockholm, Sweden
- United Kingdom (2):
  - Research Site, London
  - Research Site, Oxford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 124 subjects were screened, 22 of these were rescreened. A total of 61 subjects were assigned a treatment allocation through randomization. Two of ineligible subjects were never dispensed investigational product.
  One ineligible randomized subject was discontinued prior to dosing and refused to supply further data.
Pre-assignment Details: Protocol was administratively changed to allow reduction of sample size from 64 in this study population.
  A total of 59 completed screening and were randomized, but only 58 completed randomization and were dosed with study medication.
Groups:
- Placebo: Placebo to match AZD3241 dosed twice daily
- AZD3241 300 mg: AZD3241 300 mg dosed twice daily
- AZD3241 600 mg: AZD3241 600 mg dosed twice daily
Period: Dose Escalation Week 1
Arm/Group | Placebo | AZD3241 300 mg | AZD3241 600 mg
Started | 19 (Number randomized to treatment) | 19 (Number randomized to treatment) | 20 (Number randomized to treatment)
Completed | 17 | 16 | 18
Not Completed | 2 | 3 | 2
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Determined not eligible | 1 | 1 | 1
Period: Dose Escalation Week 2
Arm/Group | Placebo | AZD3241 300 mg | AZD3241 600 mg
Started | 17 | 16 | 18
Completed | 16 | 14 | 17
Not Completed | 1 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Determined not eligible | 1 | 1 | 1
Period: Treatment Weeks 3 to 12
Arm/Group | Placebo | AZD3241 300 mg | AZD3241 600 mg
Started | 16 | 14 | 17
Completed | 15 | 13 | 17
Not Completed | 1 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population, includes only 58 of 59 randomized subjects, those taking at least 1 dose of investigational product
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AZD3241 300 mg | AZD3241 600 mg | Total
Number analyzed (Participants) | 19 | 19 | 20 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (7.9) | 59.9 (6.1) | 58.0 (8.5) | 59 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 5 | 17
  Male | 12 | 14 | 15 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 16 | 16 | 18 | 50
  Unknown or Not Reported | 2 | 3 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 16 | 15 | 16 | 47
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 2 | 7
Multiple System Atropy Subtype [Number; unit: Participants] — Multiple System Atropy (MSA) Subtype, Parkinsonian (P) or Cerebellar (C)
  Participants
    MSA - P | 7 | 10 | 7 | 24
    MSA - C | 12 | 9 | 13 | 34
Diagnostic Category [Number; unit: Participants] — Diagnostic Category for Multiple System Atropy (MSA); Possible or Probable were the eligible categories
  Participants
    Possible MSA | 1 | 4 | 8 | 13
    Probable MSA | 18 | 15 | 12 | 45
Genotype [Number; unit: Participants] — Translocator Protein binding (TSPO) : genotype (affinity for binding); Low Affinity Binding was exclusionary
  Participants
    TSPO - High Affinity Binding | 12 | 10 | 16 | 38
    TSPO - Mixed affinity binding | 7 | 9 | 4 | 20
    TSPO- Low Affinity Binding | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Striatum Brain Region: Change From Baseline in Microglia Activation Via Positron Emission Tomography(PET)
Description: Striatum Brain region: Change from baseline in microglia activation via PET By [11C]PBR28 binding to translocator protein
Time Frame: Baseline (pre randomization) and Week 12
Population: PET analysis population (Paired baseline and week 12 PET scans)
Measure: Mean (Standard Deviation); unit: ml/cc
Arm/Group | Placebo | AZD3241 300 mg | AZD3241 600 mg
Number analyzed (Participants) | 14 | 13 | 16
ml/cc | -0.23 (0.61) | 0.12 (0.83) | -0.35 (1.25)
Statistical Analysis 1: Comparison: Placebo; Change from baseline within treatment arm; Test type: Superiority or Other; p = 0.13, ANOVA — Not adjusted; Mean Difference (Final Values) = -0.38, Standard Error of Mean 0.24 — larger negative values (powered to detect -0.50)
Statistical Analysis 2: Comparison: AZD3241 300 mg; Change from baseline; Test type: Superiority or Other; p = 0.91, ANOVA — not adjusted; Mean Difference (Final Values) = -0.03, Standard Error of Mean 0.25 — larger negative values (powered to detect -0.50)
Statistical Analysis 3: Comparison: AZD3241 600 mg; Change from baseline; Test type: Superiority or Other; p = 0.68, ANOVA; no adjustments; Mean Difference (Final Values) = -0.10, Standard Error of Mean 0.25 — larger negagtive values (powereed to detect -0.50)
Statistical Analysis 4: Comparison: Placebo vs AZD3241 300 mg; Secondary objective - comparison to placebo; Test type: Superiority or Other; p = 0.32, ANOVA — no adjustment; Mean Difference (Final Values) = 0.35, Standard Error of Mean 0.34 — Looking for negative direction to indicate treatment better than placebo
Statistical Analysis 5: Comparison: Placebo vs AZD3241 600 mg; Secondary objective; Test type: Superiority or Other; p = 0.45, ANOVA — no adjustment; Mean Difference (Final Values) = 0.28, Standard Error of Mean 0.36 — lookin for negative difference compared to placebo

2. Secondary Outcome: Myeloperoxidase (MPO) Inhibition in Plasma (Change From Baseline), Specific Activity
Description: Myeloperoxidase (MPO) inhibition in plasma (change from baseline), on samples collected and analyzed, specific activity (activity/protein)
Time Frame: Baseline (Day -1) and week 12
Population: efficacy population, restricted to subjects with paired samples analyzed within 6 months of collection
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Placebo | AZD3241 300 mg | AZD3241 600 mg
Number analyzed (Participants) | 13 | 8 | 15
ratio
  Pre dose (week 12) | 0.12 [-0.10 to 0.50] | -0.12 [-0.22 to -0.03] | -0.12 [-0.18 to -0.05]
  1 hour post dose (WEEK 12 | 0.12 [-0.30 to 0.54] | -0.10 [-0.58 to 0.39] | 0.10 [-0.27 to 0.48]
  2 to 6 hours post dose (week 12) | 0.04 [-0.04 to 0.13] | -0.15 [-0.25 to -0.08] | -0.18 [-0.26 to -0.11]

3. Other Pre Specified Outcome: Exploratory Efficacy: Unified Multiple System Atropy Rating Scale, Change From Baseline (Total Score, Part 1 + Part 2)
Description: Exploratory efficacy: Unified Multiple System Atropy Rating Scale, change from baseline (total Score, Part 1 + Part 2) : Score range 0 to 104, positive value indicates worsening symptoms
Time Frame: Baseline to final treatment visit
Population: Efficacy population: with baseline (Day -1) and post baseline assessment
Measure: Least Squares Mean (90% Confidence Interval); unit: Score change from baseline
Arm/Group | Placebo | AZD3241 300 mg | AZD3241 600 mg
Number analyzed (Participants) | 17 | 17 | 18
Score change from baseline | 4.7 [2.5 to 6.8] | 3.6 [1.4 to 5.7] | 2.6 [0.5 to 4.7]

ADVERSE EVENTS:
Time Frame: 12 weeks of randomized treation plus a follow up period up to 14 days after last dose
Description: Adverse events starting during screening period Before randomization or starting greater that 14 days after the last dose of study medication are not included in these tabulations.
Arm/Group | Placebo | AZD3241 300 mg | AZD3241 600 mg
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/19 | 1/20
Other Adverse Events (participants affected / at risk) | 14/19 | 15/19 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | AZD3241 300 mg (N=19) | AZD3241 600 mg (N=20)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Multipla System Atrophy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Subject found face down on bedding - considered disease related death
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Subject found dead with cheese in throat
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | AZD3241 300 mg (N=19) | AZD3241 600 mg (N=20)
atrial fibrilation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (3) | 3 (4)
Feeling jittery (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 2 (4) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 5 (5) | 3 (3)
Administration related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (12) | 1 (1) | 4 (6)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 1 (1)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Balance disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Clumsiness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depressive symptom (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 2 (4)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 3 (6) | 2 (4)
Hypokinesia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (2) | 2 (3)
Radicular pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Restless leg syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (4)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoe syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Alcohol use (Social circumstances) | 0 (0) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
Biomarker samples were included if testing done within 6 months of collection, recommendation changed to 3 months of collection during study. Included based on 6 months as per protocol to include as many samples as possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less